CLINICAL TRIAL: NCT05293561
Title: Cognitive Impact in Patients With COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Lecturer of Chest diseases and tuberculosis, Assiut University
Other Study IDs: WGEK-NCG
Record Dates: First submitted 2022-03-22; First posted 2022-03-24 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Cognitive Impairment; COVID-19 Respiratory Infection
Keywords: COVID-19; Cognitive Impairment; Anxiety; Depression
MeSH Terms: conditions — Cognitive Dysfunction; COVID-19; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 cases: O2 saturation readings, Mini-mental state examination (MMSE), Hamilton's anxiety (HAM-A) Hamilton's depression rating scales (HAM-D)
- control: O2 saturation readings, Mini-mental state examination (MMSE), Hamilton's anxiety (HAM-A) Hamilton's depression rating scales (HAM-D)

SUMMARY:
SARS-COV-2 (severe acute respiratory syndrome- corona virus - 2) infection reframed medical knowledge in many aspects, yet there is still a lot to be discovered. Coronavirus disease 19 (COVID-19) can cause neuropsychiatric, psychological and psychosocial impairments. Literature regarding cognitive impact of COVID-19 is still limited.

Objective: evaluation of cognitive function, anxiety and depression among patients with Coronavirus disease 19.

DETAILED DESCRIPTION:
COVID-19 results in a variety of symptoms with multi-organ affection, including fever, cough; grave respiratory symptoms, gastrointestinal manifestations and fatigue. As more is learned, neurological and psychological symptoms appear to manifest in a large subscale of patients. Headache, dizziness and even a cerebrovascular event have been reported. Anosmia and ageusia reported as early indicators of SARS-CoV-2 infection, suggesting that early neurological involvement may be relevant.

Public health emergencies as COVID-19 are likely to cause adverse neuropsychiatric impacts. Cognitive impairments after SARS-COV-2 infection were noticed, COVID-19 patients complain of poor concentration, declined memory, and insomnia, as well as anxiety and depression symptoms.

The battle against COVID-19 is still continuing worldwide. People's adherence to confinement regulations and response to vaccination campaigns is essential, which is largely affected by their knowledge, attitudes, and practices towards COVID-19. Home isolation and social distancing are also associated with fear, frustrations, uncertainty, anxiety and depressive symptoms.

During the acute phase of COVID-19 infection, about 36% of cases develop neurological symptoms of which 25% can be attributed to the direct involvement of the central nervous system. Patients who show neurological symptoms included cases with or without pre-existing neurological disorders. While on intensive care units, patients showed agitation, confusion, and corticospinal tract signs such as enhanced tendon reflexes and clonus. COVID-19 can further lead to changes of coagulation and, in particular, to inflammation-induced disseminated intravascular coagulation (DIC).

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients diagnosed using Real Time-Polymerase Chain Reaction to confirm the diagnosis

Exclusion Criteria:

* neurological disorders, psychological disorders, dementia, Alzheimer's disease, end-organ failure conditions

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients diagnosed using Real Time-Polymerase Chain Reaction to confirm the diagnosis and healthy control belonging to either gender. COVID-19 patients recruited from home isolation at first visit in outpatient clinic and then after end of isolation period for 14 days, patients included from hospital isolation ward; also recruited from the respiratory isolation ICU, chest department of Assiut university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Cognitive impairment | 1 month
  degree of affection in cognition due to COVID-19 infection

SECONDARY OUTCOMES:
Level of Anxiety and depression among COVID-19 cases | 1 month
  Level of Anxiety and depression among COVID-19 cases

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Gamal elddin, MD, Principal Investigator — Assiut university hospitals
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alemanno F, Houdayer E, Parma A, Spina A, Del Forno A, Scatolini A, Angelone S, Brugliera L, Tettamanti A, Beretta L, Iannaccone S. COVID-19 cognitive deficits after respiratory assistance in the subacute phase: A COVID-rehabilitation unit experience. PLoS One. 2021 Feb 8;16(2):e0246590. doi: 10.1371/journal.pone.0246590. eCollection 2021. PMID 33556127
- [Background] Germani A, Buratta L, Delvecchio E, Gizzi G, Mazzeschi C. Anxiety Severity, Perceived Risk of COVID-19 and Individual Functioning in Emerging Adults Facing the Pandemic. Front Psychol. 2020 Dec 7;11:567505. doi: 10.3389/fpsyg.2020.567505. eCollection 2020. PMID 33364996